CLINICAL TRIAL: NCT05037266
Title: Cohort Assessing the Immunogenicity and the Safety of the COVID-19 Vaccine Janssen in Healthy Volunteers Based on 2 Age Groups: 65 Years or Older - 55 to 65 Years. Covicompare-Janssen
Acronym: CoviCompare_J
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was stopped due to lack of inclusions
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21CH135; 2021-003191-14 (EudraCT Number)
Record Dates: First submitted 2021-09-06; First posted 2021-09-08 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Healthy Volunteers
Keywords: vaccine; immunity; immunogenicity; Janssen vaccine; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Ad26COVS1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 55 - 64 years old (50 volunteers) (Experimental): 1 injection of vaccine Janssen (Ad26.COV2-S) at Day 1 and boost vaccine at Day 57
  Interventions: Biological: COVID-19 Vaccine Janssen (Ad26.COV2-S)
- At least 65 years old (50 volunteers) (Experimental): 1 injection of vaccine Janssen (Ad26.COV2-S) at Day 1 and boost vaccine at Day 57
  Interventions: Biological: COVID-19 Vaccine Janssen (Ad26.COV2-S)

INTERVENTIONS:
Biological: COVID-19 Vaccine Janssen (Ad26.COV2-S) — one dose (0.5mL) at D1 and one dose (0.5mL) at D57

SUMMARY:
In response to the COVID-19 pandemic, several vaccines (Pfizer, Moderna, Astrazeneca, Janssen) have been developed and are being administered to millions of people in France and billions around the world through massive vaccination programs.

The Janssen vaccine is the fourth COVID-19 vaccine to be licensed in Europe. It received a European marketing authorization for all adults, without age limit, on March 11, 2021. Janssen's vaccine is a viral non replicating vector (adenovirus) vaccine targeting the Spike protein of the SARS-CoV-2 virus. It differs from currently available vaccines in that it is a single-dose regimen with significant protection at 28 days post-injection. Monitoring of the durability of the immune response is essential to assess the need for a booster vaccination. Insufficient data are available in the adult population regarding the evolution of the immune response. This point seems to be even more important in the elderly. Indeed, their immune system declines with age, leading to a greater susceptibility to infectious diseases and a weaker response to vaccination. This is called immunosenescence. Vaccination in this population is essential to avoid severe COVID-19 cases, since older people are particularly at risk.

Two CoviCompare studies with two licensed vaccines messenger RNA vaccines (Pfizer, Moderna) are underway to evaluate the immune response to each vaccine according to age.

We propose to conduct a study to evaluate the immunogenicity of the Janssen vaccine in different age groups with long-term follow-up. This will allow determining the need of a booster.

A common battery of in vitro and ex vivo immuno-monitoring tests has been set up to systematically assess the acquisition of humoral and cellular immunity over time over a period of 24 months following vaccination in the CoviCompare project. This trial, part of the CoviCompare project will use the same immunomonitoring set. This will also allow comparison of the immune response to different vaccines in subjects of different age in order to determine in this at risk population the better vaccination schedules.

The only difference between this trial and the other 2 trials of the CoviCompare project is that adults aged 18-45 will not be concerned here, because the adenovirus vaccine is not recommended for this age group in France

DETAILED DESCRIPTION:
In this trial of the Covicompare project, we will therefore evaluate the immune response after Janssen vaccine in subjects aged more than 65 years and 55 to 65 years without a prior COVID-19, following the same immunomonitoring analyses as for the other CoviCompare project trials.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults, or stable medical condition for adults with pre-existing medical conditions. A stable medical condition is defined as disease not requiring significant change in therapy or hospitalization for worsening disease during 3 months before enrolment, nor expected to require any significant change in therapy or hospitalization for worsening disease in foreseeable future.
* Understands and agrees to comply with the study procedures (visits, phone calls) and provides written free informed consent.
* Able to comply with study procedures based on Investigator judgement.
* Affiliated to a social security system, (except state medical aid)

Exclusion Criteria:

* Subject is ill or febrile (body temperature ≥ 38.0°C) within 72 prior hours or and/or symptoms suggestive of COVID-19 within the past 14 days at enrolment visit (ill or febrile participants may be re-scheduled within the inclusion period when no longer presenting symptoms)
* History of documented COVID-19 (PCR+, antigenic test+ or chest CT Scan + or serology SARS-CoV- 2+) prior to the vaccine administration
* Subjects with positive serology to SARS-CoV-2 at the enrolment visit.
* Subjects who already received another anti-SARS-CoV-2-vaccine
* Subjects who received BCG (Bacille Calmette and Guérin vaccine) given within the last year.
* An immediate family member or household member of study staff.
* Use of immunosuppressive drugs like e.g. corticosteroids at a dosage > 10mg/day (excluding topical preparations and inhalers) within 3 months prior to enrolment or 6 months for chemotherapies
* Received immunoglobulin or other blood product within 3 months prior to enrolment or planned receipt of immunoglobulin or a blood product through study completion.
* Received any vaccination within 4 weeks prior to first injection or plan to receive a licensed vaccine 4 weeks after the last injection (exception for flu vaccine within 2 weeks).
* History of severe adverse reactions to vaccine administration, including anaphylaxis and related symptoms, such as rash, respiratory difficulty, angioedema and abdominal pain to vaccines, or history of allergic reaction likely to be exacerbated by any component of the anti-SARS-CoV-2- vaccine.
* History of severe allergic event
* Participation in another investigational clinical study within 4 weeks before the enrolment visits or planned before the study completion.
* Known HIV (human immunodeficiency virus), active HCV (Hepatitis C virus) or HBV (Hepatitis B virus) infection
* Any pathological condition, such as cancer, which may be susceptible of reducing immunity response
* History of heparin-induced thrombocytopenia (HIT)
* Any bleeding disorder considered as contraindication to intramuscular injection or phlebotomy
* The use of investigational Ig, investigational monoclonal antibodies or convalescent serum are not allowed during the study
* Any condition which in the opinion of the investigator may interfere with the aim of the study
* Pregnant or breastfeeding or positive pregnancy urine test at enrolment visit.
* Woman in childbearing without efficacious contraception (in the opinion of the investigator) for 31 days after treatment
* People under legal protection measure (tutorship, curatorship or safeguard measures)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
IgG humoral response to vaccine | Day 29
  Anti SARS-CoV-2 Spike IgG as measured by ELISA

SECONDARY OUTCOMES:
IgG humoral response to vaccine | Day 1, Day 29, Day 57, Month 6, Month 12, Month 24
  Anti SARS-CoV-2 Spike IgG (total and subclasses IgG 1-4) as measured by ELISA
IgA humoral response to vaccine | Day 1, day 29, Day 57, Month 6, Month 12, Month 24
  Anti SARS-CoV-2 Spike IgA as measured by Elisa
IgM humoral response to vaccine | Day 1, day 29, Day 57, Month 6, Month 12, Month 24
  Anti SARS-CoV-2 Spike IgM as measured by Elisa
neutralizing antibody humoral response to vaccine | Day 1, day 29, Day 57, Month 6, Month 12, Month 24
  Anti-SARS-CoV-2 neutralizing antibody (pseudo-neutralization test using lentiviral models expressing SARS-Cov-2 proteins)
T cells response to vaccine | Day 1, Day 57, Month 6
  Fluorospot assays (TH1, TH2, TH17, Cytotoxicity). Phenotyping of SARS-CoV-2 specific T cells by mass cytometry
Mucosal response to vaccine | Day 1, day 29, Day 57, Month 6, Month 12, Month 24
  Mucosal SARS-CoV-2 -specific antibody via measure of sIgA, sIgM and IgG in saliva by specific home-made and commercially available ELISA assays.
B cell response to vaccine | Day 1, Day 57, Month 6
  Determination of the epitope profiling and B cell repertoire (stereotype clonotype) of the humoral response

CONTACTS AND LOCATIONS:
Overall Officials: ELISABETH BOTELHO-NEVERS, MDPHD, Principal Investigator — CENTRE HOSPITALIER DE SAINT-ETIENNE
Locations (10):
- France (10):
  - Chu de Dijon, Dijon
  - Centre Hospitalier Regional Lille, Lille
  - APHM, Marseille
  - Centre Hospitalier Universitaire Nantes, Nantes
  - Hopital Bichat, Paris
  - Hopital Cochin, Paris
  - Centre Hospitalier Universitaire Rennes, Rennes
  - Chu de Rouen, Rouen
  - Centre Hospitalier de Saint-Etienne, Saint-Etienne
  - Centre Hospitalier Tours, Tours

IPD SHARING:
Plan to Share IPD: No